CLINICAL TRIAL: NCT02329067
Title: The Metabolic Effect of Walnut Consumption in Healthy Men and Healthy Postmenopausal Women Substituting Walnuts for Different Food Components
Brief Title: The Metabolic Effect of Walnuts in Healthy Subjects
Acronym: WALDI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Klaus Parhofer, professor of Endocrinology and Metabolism, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: WALNUT-2
Record Dates: First submitted 2014-12-29; First posted 2014-12-31 (Estimated); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Lipid Metabolism Disorders
MeSH Terms: conditions — Lipid Metabolism Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- walnut-CH (Experimental): Western type diet including walnuts (43g/day); Walnuts substitute carbohydrates
  Interventions: Other: walnuts
- Walnut-SFA (Experimental): Western type diet including walnuts (43g/day); Walnuts substitute saturated fatty acids
  Interventions: Other: walnuts
- Walnut-LIB (Experimental): Western type diet including walnuts (43g/day); no specific recommendation
  Interventions: Other: walnuts
- Control (No Intervention): Isocaloric western type diet w/o nuts, nut butters or nut oils of any kind

INTERVENTIONS:
Other: walnuts — consumption of 43 g walnuts per day
  Arms: Walnut-LIB; Walnut-SFA; walnut-CH

SUMMARY:
The objectives of the proposed study are to assess whether the metabolic effects of walnut consumption depends on which food components the walnuts substitute (i.e. carbohydrates; saturated fatty acids) and whether it is important to consume walnuts as snacks or with meals.

DETAILED DESCRIPTION:
The objectives of the proposed study are to assess whether the metabolic effects of walnut consumption depends on which food components the walnuts substitute (i.e. carbohydrates; saturated fatty acids) and whether it is important to consume walnuts as snacks or with meals.

The metabolic effects of walnut consumption may not only relate to the ingested walnuts but also to what is not eaten when walnuts are consumed. We want to evaluate whether the metabolic changes are more pronounced if study participants are instructed to reduce carbohydrates or saturated fatty acids to remain on an isocaloric diet. In a third group we will test what food is omitted if no specific instructions are given. Furthermore half of the subjects in each group will be instructed to eat walnuts with meals and half as snacks.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal healthy women and healthy men
* Age >50 yrs
* Written informed consent prior to study participation

Exclusion Criteria:

* Known allergy to nuts
* Evidence of alcohol (women >70g/week, men >140g/week), tabacco or drug abuse
* Obesity ≥35 kg/m2
* Diabetes mellitus
* Hypertension >140/90 mmHg or history of hypertension
* LDL-cholesterol >190 mg/dl, Triglycerides > 350 mg/dl
* History of atherosclerotic disease
* Liver disease of any etiology
* Kidney disease of any etiology (GFR < 60 ml/min/1.73)
* Uncontrolled thyroid disease or other endocrine diseases
* Acute or chronic inflammatory diseases
* Active malignancy
* Current or previous (within 3 months) treatment with antidiabetic drugs, hypolipidemic drugs, antihypertensive drugs, anti-inflammatory drugs, vitamin E, hormonal replacement therapy
* major surgical intervention within 3 months (or planned)

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2014-12; Primary Completion 2016-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Non-HDL-cholesterol | 8 weeks

SECONDARY OUTCOMES:
LDL-cholesterol | 8 weeks
total-cholesterol | 8 weeks
apoB | 8 weeks
triglycerides | 8 weeks
fasting glucose | 8 weeks
HOMA index | 8 weeks
caloric intake | 8 weeks
ratio CH:fat:protein | 8 weeks
ratio SFA:MUFA:PUFA | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Klaus G Parhofer, MD, Principal Investigator — Ludwig-Maximilians - University of Munich
Locations (1):
- Medical Department 2, University Munich, Munich, Germany